CLINICAL TRIAL: NCT07235904
Title: Efficacy of Top-down Therapy With Mirikizumab Versus Standard of Care With Azathioprine in Patients With Newly Diagnosed Moderate-to-severe Ulcerative Colitis: A 52-week, Multicenter, Open-label, Randomized Controlled Trial
Brief Title: Efficacy of Top-down Therapy With Mirikizumab Versus Standard of Care With Azathioprine in Patients With Newly Diagnosed Moderate-to-severe Ulcerative Colitis
Acronym: MIRACLE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRACLE; 2025-522585-72-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-30; First posted 2025-11-19 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirikizumab (Experimental)
  Interventions: Drug: Mirikizumab
- Azathioprine (Active Comparator)
  Interventions: Drug: Azathioprine (AZA)

INTERVENTIONS:
Drug: Mirikizumab — Patients in the mirikizumab arm will receive an initial 300 mg dose every 4 weeks intravenously for three doses during the 12-week induction period.After completing induction, patients will switch to maintenance therapy with 200 mg mirikizumab subcutaneously.
  Arms: Mirikizumab
Drug: Azathioprine (AZA) — Patients in the azathioprine arm will receive oral azathioprine at a dose of 2.0-2.5 mg/kg body weight daily in combination with an initial daily dose of 40-60 mg glucocorticoids, which may be tapered as clinically appropriate.
  Arms: Azathioprine

SUMMARY:
The MIRACLE trial is for patients who have been newly diagnosed with moderate to severe ulcerative colitis in the last 12 months and who have not responded adequately to treatment with mesalazine and prednisolone alone. The standard drug therapy for ulcerative colitis begins with mesalazine (+cortisone) and, if the response is insufficient, continues with azathioprine (+cortisone). Only in the next step are biologics (biotechnologically produced protein substances such as antibodies) such as mirikizumab used as needed. Recent studies have now shown that earlier treatment with mirikizumab without prior treatment with azathioprine may be more effective in the long term, and there are indications that this may result in fewer side effects. This study aims to investigate whether direct, early treatment with mirikizumab is more effective than the usual initiation of standard therapy with azathioprine, whereby these patients can then switch to mirikizumab at predetermined times during the course of the study from week 24 onwards if they have a defined disease activity despite the previous azathioprine treatment. The study consists of an initial treatment period of 12 weeks (induction therapy) and a maintenance therapy period of 40 weeks. Patients in the mirikizumab arm receive 12 doses of mirikizumab. This includes initially 300 mg intravenously every 4 weeks at the trial site, followed by 200 mg subcutaneously via two subcutaneous injections of 100 mg each, administered independently at home. In the azathioprine arm patients receive daily administration of azathioprine tablets in combination with a steroid. Assignment to one of the two treatment options is randomised with equal probability for each of the treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent prior to any study-specific procedures being completed.
2. Are willing and able to complete the scheduled study assessments, including endoscopy and daily diary entry.
3. Are willing to comply with contraception requirements (as specified in section 7.7)
4. Age between 18 and 75 years.
5. Naïve to azathioprine and its metabolite 6-MP
6. Naïve to advanced therapies.
7. Early disease (duration < 12 months since first diagnosis).
8. Patients with active ulcerative colitis (UC) for whom a previous therapy with 5-aminosalicylic acid (5-ASA) or steroids have not worked well enough, have stopped working, or have caused unacceptable side effects.
9. The steroid oral therapy must have been stable for at least two weeks before baseline and may consist of prednisone ≤20 mg/day (or equivalent) per os.
10. The oral 5-ASA therapy must have been ongoing for at least 8 weeks and dose must be stable for at least 2 weeks before baseline.
11. Modified Mayo score (mMS) 5-9.
12. Endoscopic Mayo (eMayo) score ≥2 (local).
13. Robarts Histopathology Index (RHI) >4 (central)
14. Elevated CRP (above the upper limit of normal) or Fcal (above 250 ug/g stool).
15. Disease localization involving at least the rectum and sigmoid colon (>15 cm).

Exclusion Criteria:

1. Fulminant ulcerative colitis patients who do not respond to steroid treatment or requiring >20 mg of prednisolone (or equivalent) at baseline and/or fulfilling the criteria for severe UC (requirement of hospitalization) .
2. Patients with complex UC who have required cyclosporine and tacrolimus for previous treatment
3. Treatment with MTX within 8 weeks before baseline
4. Rectal 5-ASA or rectal steroids treatment within 2 weeks prior to baseline
5. History of malignancy, except for non-melanoma skin cancer.
6. Planned or foreseeable surgery at the time of inclusion.
7. Known thiopurine methyltransferase deficiency.
8. Known hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption.
9. Diagnosis of Crohn's disease.
10. Have been diagnosed with clinically important infection including, but not limited to, hepatitis B, hepatitis C, HIV/AIDS, and active tuberculosis (TB).
11. Have detectable hepatitis B virus (HBV) DNA. or hepatitis C virus (HCV) RNA
12. Have been diagnosed with latent TB and are not willing to comply with completing TB treatment as appropriate.
13. Intend to receive a Bacillus Calmette-Guerin (BCG) vaccination or live attenuated vaccine(s) during the study.
14. Have been diagnosed with systemic mycoses and parasitosis
15. Have an unstable or uncontrolled illness, including, but not limited to, cerebrocardiovascular, respiratory, gastrointestinal (excluding UC), hepatic, renal, endocrine, hematologic or neurological disorders or malignancy that would potentially affect patient safety within the study or confound efficacy assessment.
16. Have a known systemic hypersensitivity to any component of this investigational product or has experienced an acute systemic hypersensitivity event with previous study drug administration, that precludes mirikizumab therapy.
17. Women who are pregnant, lactating or planning pregnancy
18. Became a Lilly employee or employee of any of the organizations involved with this study or study site personnel directly affiliated with this study and/or their immediate families.
19. Have participated in another clinical trial involving an investigational product or nonapproved use of a drug during the last twelve weeks before screening or are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
20. Are unwilling or unable to comply with the use of a data collection device to directly record data from the patient daily for the duration of Study MIRACLE or are unable to complete other study procedures.
21. Have been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
comprehensive disease control | Week 52
  The proportion of patients achieving comprehensive disease control at Week 52, defined as: Steroid-free clinical remission (modified Mayo score remission [ES ≤1, SF ≤1, RB=0] and no glucocorticoid use for at least 12 weeks prior to week 52) achieved without surgery, and Biochemical remission (CRP <0.5 mg/dl and Fcal <250 μg/g stool), and Endoscopic improvement (eMayo=0-1), and Histologic remission (RHI ≤3, with subscores of 0 for lamina propria neutrophils and of 0 for neutrophils in epithelium), and Normalization of IBD-related QoL (sIBDQ ≥60 points).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Schleswig-Holstein, Kiel, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data resulting from the MIRACLE trial will be made available upon request under the following pre-requisites: Only data from already published results will be made available to academic researchers upon reasonable request, e.g. for meta-analyses. Data will be shared after deidentification in an aggregated form. This requires approval by the local Institutional Review Board of the researcher requesting the data in advance.